CLINICAL TRIAL: NCT06318702
Title: The Effect of Constructivist Learning Model Based Gynecological Cancer Education on Gynecologic Cancer Awareness, Spiritual Well-being and Health Anxiety: A Randomized Controlled Trial
Brief Title: The Effect of Constructivist Learning Model Based Gynecological Cancer Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Şahika ŞİMŞEK ÇETİNKAYA, Head of Midwifery, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2023-KAEK-180
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Gynecologic Cancer
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KETEM (No Intervention): This group was given a three-week standard gynecological cancer education program by the Cancer Early Diagnosis, Screening and Education Centers (KETEM) unit.
- constructivist model group (Experimental): Gynecologic cancer education was given to the intervention group for 3 weeks based on the constructivist education model, taking into account the assimilation, adaptation and balancing stages of education.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — is an education program implemented to raise women's awareness about reproductive health and to help them adopt healthy habits.
  Arms: constructivist model group

SUMMARY:
This is a randomised controlled study.The study was conducted to determine the effect of the constructivist education model given to women on gynecological cancer awareness, health Anxiety and spiritual well-being in women . The study population was composed of women living in Kastamonu. Women will be assigned to control and experimental groups. Women in the control group will receive gynecological education from Cancer Early Diagnosis, Screening and Education Centers (KETEM). The other group will receive gynecological cancer education based on the constructivist model.The hypotheses of the study are as follows:

H0: The of constructivist learning model -based health education programme does not have an effect on gynecologic cancer awareness, spiritual well-being and health anxiety.

H1: The of constructivist learning model -based health education programme have an effect on gynecologic cancer awareness, spiritual well-being and health anxiety.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years old,
* being willing to participate in this study

Exclusion Criteria:

* having any neuropsychiatric disorder,
* having any physical or mental illness,
* being diagnosed with gynecological cancer,
* not attending theoretical trainings.

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-12-25 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
gynecologic cancer awareness | before education, after education, 4 weeks after education
  comparing the two groups in terms of gynecologic cancer awareness scores. Gynaecological cancer awareness scale will use for data collecting. This scale consists of 41 items and four sub-dimensions, with a minimum score of 41 and a maximum score of 205.The awareness of women is greater the higher the scores obtained from the scale.
spiritual well-being | before education, after education, 4 weeks after education
  comparing the two groups in terms of spiritual well-being scores.Three-Factor Spiritual Well-Being Scale will use for collecting data.The scale is graded on a 5-point Likert scale (1=Not at all appropriate for me, 2=Not appropriate for me, 3=A little appropriate for me, 4=Quite appropriate for me, 5=Exactly appropriate for me). . An increase in the score obtained from the scale indicates an increase in the spiritual well-being of the individual
health anxiety scores | before education, after education, 4 weeks after education
  comparison of the two groups in terms of health anxiety scores.Health Anxiety Inventory will use for data collecting.. It is an 18-item self-report inventory. Each item is scored from 0 to 3 The maximum score that can be obtained from the scale is 54 and higher scores indicate higher levels of HAI

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Merkez, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No